CLINICAL TRIAL: NCT03250091
Title: Surveillance Strategies of Patients With Precancerous Conditions and Lesions in the Stomach
Brief Title: Surveillance of Patients With Precancerous Lesions of the Stomach
Status: Recruiting | Type: Observational
Sponsor: University of Latvia (Other)
Collaborators: Digestive Diseases Centre GASTRO (Other); Riga East Clinical University Hospital (Other Government); Academic Histology Laboratory (Latvia) (Other)
Responsible Party: Sponsor
Other Study IDs: 2915
Record Dates: First submitted 2017-07-21; First posted 2017-08-15 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Gastric Cancer; Gastric Intestinal Metaplasia; Gastric Atrophy; Gastric Dysplasia
Keywords: gastric precancerous lesions; gastric cancer; gastric intestinal Metaplasia; gastric atrophy; gastric dysplasia
MeSH Terms: conditions — Stomach Neoplasms; Gastritis, Atrophic | interventions — Gastroscopy; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human biopsy samples that are used for histopathology analysis are containing human DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Gastric cancer: Gastric adenocarcinoma and other gastric malignancies
  Interventions: Procedure: Upper endoscopy with biopsies; Procedure: Plasma/serum sampling; Procedure: Biopsies for gastric microbiota; Procedure: Faecal sample acquisition
- Gastric mucosal dysplasia: Includes: a. High-grade dysplasia; b. Low-grade dysplasia; c. Indefinite for dysplasia
  Interventions: Procedure: Upper endoscopy with biopsies; Procedure: Plasma/serum sampling; Procedure: Biopsies for gastric microbiota; Procedure: Faecal sample acquisition
- High-risk IM gastritis stages: High-risk stages according to OLGIM classification: OLGIM Stage IV and OLGIM Stage III.
  Interventions: Procedure: Upper endoscopy with biopsies; Procedure: Plasma/serum sampling; Procedure: Biopsies for gastric microbiota; Procedure: Faecal sample acquisition
- High-risk atrophic gastritis stages: High-risk stages according to OLGA classification: OLGA Stage IV and OLGA Stage III.
  Interventions: Procedure: Upper endoscopy with biopsies; Procedure: Plasma/serum sampling; Procedure: Biopsies for gastric microbiota; Procedure: Faecal sample acquisition
- Extensive gastric intestinal metaplasia: Intestinal metaplasia of any grade both in gastric corpus and antrum/incisura (other than OLGIM III-IV).
  Interventions: Procedure: Upper endoscopy with biopsies; Procedure: Plasma/serum sampling; Procedure: Biopsies for gastric microbiota; Procedure: Faecal sample acquisition
- Extensive atrophy: Moderate to severe (++ or +++) atrophy both in corpus and antrum/incisura, other than OLGA III-IV.
  Interventions: Procedure: Upper endoscopy with biopsies; Procedure: Plasma/serum sampling; Procedure: Biopsies for gastric microbiota; Procedure: Faecal sample acquisition
- Isolated corpus atrophy: Isolated moderate-to-severe atrophy or IM in the corpus.
  Interventions: Procedure: Upper endoscopy with biopsies; Procedure: Plasma/serum sampling; Procedure: Biopsies for gastric microbiota; Procedure: Faecal sample acquisition

INTERVENTIONS:
Procedure: Upper endoscopy with biopsies — Upper endoscopy with proper biopsy work-up will be used for identification and stratification of gastric lesions as well as acquisition of biopsies for histopathological examination, including H.pylori detection
  Other Names: gastroscopy, upper endoscopy
Procedure: Plasma/serum sampling — Plasma/serum sampling will be used to obtain information for group stratification, e.g. H.pylori status determination, serum biomarkers
Procedure: Biopsies for gastric microbiota — During upper endoscopy biopsies for gastric microbiota analysis will be obtained
Procedure: Faecal sample acquisition — Faecal samples will be obtained for faecal occult blood testing as well as microbiota analysis

SUMMARY:
The project will aim to identify and determine subgroups of patients with different risks of progression to gastric cancer and to assess appropriate follow-up intervals. Implementing risk stratification only high risk individuals will be offered and performed endoscopic surveillance.

DETAILED DESCRIPTION:
Gastric cancer is still an important healthcare problem with significant mortality rates. Latvia is a high incidence country of gastric cancer. Unfortunately most of the gastric cancer cases in Latvia are diagnosed at late stages when the treatment is substantially less effective.

Ideally, gastric cancer could be prevented by detecting gastric precancerous conditions/lesions and identifying those individuals at high-risk of progressing to cancer to the follow-up.

Population based endoscopic screening for gastric cancer is not recommended for the early detection of gastric cancer generally deemed not to be cost-effective.

However, in the absence of screening, patients present with advanced disease, and prognosis is poor.

Targeted endoscopic surveillance strategies for gastric cancer should be introduced following the principles of the recent European guidelines: Management of precancerous conditions and lesions in the stomach (MAPS) (Dinis-Ribeiro, Areia et al. 2012).

The project will aim to identify and determine subgroups of patients with different risks of progression to gastric cancer and to assess appropriate follow-up intervals. Implementing risk stratification only high risk individuals will be offered endoscopic surveillance.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing upper endoscopy Motivation to participate in the study Signed consent

Exclusion Criteria:

Known gastric cancer Unwillingness or inability to co-operate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients with material of standardized biopsies according to the standard criteria (updated Sydney system) will be classified in different risk groups for progression to gastric cancer (Group 2-7).
  The appropriate follow-up intervals will be scheduled according MAPS guidelines and follow-up procedures (upper endoscopies) will be performed for each research group (Group 2-7).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-06-19 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Risk stratification | At baseline
  The patients with material of standardized biopsies according to the standard criteria (updated Sydney system) will be classified in different risk groups for progressing to gastric cancer.
  The measurements for the risk stratification will be used following the updated Sydney grading and classification system e.g. degree and extent of atrophy, intestinal metaplasia and dysplasia in the stomach mucosa

SECONDARY OUTCOMES:
Scheduled follow-up procedures (gastroscopies) for high risk group patients | At baseline and then 1 and 3 years after the intervention depending on hystopathological report through study completion
  The subgroup of patients at different risk of progression to gastric cancer will be selected and appropriate follow-up intervals will be scheduled and performed. Significant risk stage changes before and after the follow-up upper endoscopy in different research groups.
Gastric, faecal microbiome in cancer patients and patients with precancerous lesions | At baseline and then 1 and 3 years after the intervention depending on hystopathological report through study completion
  Significant differences in the composition of gastric, faecal microbiome (phyla, genera) in cancer patients and patients with precancerous lesions

CONTACTS AND LOCATIONS:
Overall Officials: Marcis Leja, Prof.,PhD, Study Director — Institute of Clinical and Preventive Medicine, University of Latvia
Locations (1):
- University of Latvia, Riga, Latvia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dinis-Ribeiro M, Areia M, de Vries AC, Marcos-Pinto R, Monteiro-Soares M, O'Connor A, Pereira C, Pimentel-Nunes P, Correia R, Ensari A, Dumonceau JM, Machado JC, Macedo G, Malfertheiner P, Matysiak-Budnik T, Megraud F, Miki K, O'Morain C, Peek RM, Ponchon T, Ristimaki A, Rembacken B, Carneiro F, Kuipers EJ; European Society of Gastrointestinal Endoscopy; European Helicobacter Study Group; European Society of Pathology; Sociedade Portuguesa de Endoscopia Digestiva. Management of precancerous conditions and lesions in the stomach (MAPS): guideline from the European Society of Gastrointestinal Endoscopy (ESGE), European Helicobacter Study Group (EHSG), European Society of Pathology (ESP), and the Sociedade Portuguesa de Endoscopia Digestiva (SPED). Endoscopy. 2012 Jan;44(1):74-94. doi: 10.1055/s-0031-1291491. Epub 2011 Dec 23. PMID 22198778